CLINICAL TRIAL: NCT04046315
Title: Early Detection of Cardiac Damage With CMR in Women With Breast Cancer
Acronym: EARLY-CATCH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 108818
Record Dates: First submitted 2019-08-01; First posted 2019-08-06 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2019-08

CONDITIONS: Cardiotoxicity; Breast Cancer; Chemotherapy Induced Systolic Dysfunction
MeSH Terms: conditions — Cardiotoxicity; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CMR — GLS measurement with CMR

SUMMARY:
With this study the investigators will assess early cardiac damage by means of Global Longitudinal Strain (GLS) in newly diagnosed breast cancer (BC) patients treated with anthracycline-based chemotherapy, and to investigate whether myocardial damage as measured with T1 / T2 Cardiovascular Magnetic Resonance (CMR) mapping and plasma hs-Troponin T is related to changes in GLS.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age ≥ 18 years
* A diagnosis of primary breast cancer
* Starting (neo-) adjuvant chemotherapy treatment within 2 months after screening
* Cardiotoxicity risk score of intermediate, high or very high risk

Exclusion Criteria:

* Previous radiotherapy or systemic cancer treatment
* Cancer metastasis
* Life expectancy of less than 6 months
* History of myocardial infarction or heart failure
* Known contra-indications for CMR
* Refusal or inability to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be recruited from the general BC population receiving (neo-) adjuvant chemotherapy. Patients with a new diagnosis of malignant neoplasm of the breast, codes C50.0-C50.9, according to the World Health Organization International Classification of Diseases (WHO-ICD) will be eligible for participation.
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Global Longitudinal Strain (GLS) change after chemotherapy compared to baseline | Baseline and 2 weeks after the last chemotherapy cycle
  A relative reduction in Global Longitudinal Strain (GLS) assessed with CMR

CONTACTS AND LOCATIONS:
Overall Officials: Saloua El Messaoudi, PhD, Study Chair — Radboud University Medical Center; Angela Maas, PhD, Principal Investigator — Radboud University Medical Center; Robin Nijveldt, PhD, Study Chair — Radboud University Medical Center
Locations (1):
- Radboud University Medical Center, Nijmegen, Netherlands